CLINICAL TRIAL: NCT04463524
Title: Screening of Patients With Suspected Heart Rhythm Disorder on Primary Health Care Level With the Use of Personal Digital ECG Sensor
Brief Title: Screening for Hearth Rhythm Disorders
Status: Completed | Type: Observational
Sponsor: Healthcare Center Murska Sobota (Other)
Responsible Party: Principal Investigator, Stasa Vodicka, asist. prof. Stasa Vodicka, MD, Healthcare Center Murska Sobota
Other Study IDs: UESVADZ001
Record Dates: First submitted 2020-06-22; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Arrhythmia
Keywords: Heart rhythm disorder; palpitation; primary healthcare; personal mobile ECG sensor; referral
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test: They will receive ECG sensor after initial standard 12-channel ECG record will be taken; they will return after 5 days and after 3 months to assess their hearth rhythm disorders and actions taken.
  Interventions: Device: Personal ECG digital sensor
- Control: They will not receive ECG sensor after initial standard 12-channel ECG record will be taken; they will return after 5 days and after 3 months to assess their hearth rhythm disorders and actions taken.
  Interventions: Device: Personal ECG digital sensor

INTERVENTIONS:
Device: Personal ECG digital sensor — Patients in test group will receive personal ECG sensor and in control gropu will not.
  Other Names: Savvy Personal ECG digital sensor

SUMMARY:
This study aimed to analyze the usefulness of telecardiology in the primary health care level using an ECG personal sensor developed in Slovenia.Investigators also wanted to evaluate the satisfaction of patients and their physicians and the cost-effectiveness of this tool.

DETAILED DESCRIPTION:
This observational prospective cohort study was conducted on patients with a history of rhythm disturbance who visited their family physician at the Health Care Center of Ljubljana and Health Care Center of Murska Sobota from October 2016 to January 2018. It included family physicians and their patients and was conducted on two levels. The inclusion criteria were age of ≥18 years, suspected heart rhythm disorder, and no previous diagnosis of rhythm disorder. Patients had a 12-channel ECG record performed at the first visit. If a rhythm disturbance was detected at that time, the patient was treated according to the guidelines and was not included in the study. However, if a diagnosis of rhythm disorder could not have been made, the patient was included in the study. In the study, the investigators divided participants into two groups: the test group and control group, where the patients in the test group received a wearable device. The pilot study is a part of an ongoing study that includes a bigger sample calculated with the help of Raosoft sample size calculator. Investigators estimated that a sample size of 100 patients (50 in test and 50 in the control group) is sufficient to obtain relevant data in the population. Patients who met these criteria were invited to participate in a study that was approved by the Ethics Committee of the Republic of Slovenia (number 0120-299/2017-7, KME 47/06/17), and written informed consent confirmed their participation. The study was conducted in accordance with The Code of Ethics of the World Medical Association (Declaration of Helsinki).

In collaboration with medical experts, the Jožef Stefan Institute of Slovenia developed a personal portable ECG sensor that works in conjunction with a smartphone. The Personal Digital Mobile Body Sensor is listed in the medical device category, has the status of a medical device with all necessary certifications, and is owned by Savvy. It includes a personal sensor, ECG electrode kit, MobECG mobile application, and computer program called VisECG, which is currently available for Android only. The ECG sensor consists of two electrodes, which are placed 8.5 cm apart, and measures the potential between these two closely placed body-surface electrodes. The gadget weighs 21 g and has several possible positions of placement. The measurement is transmitted via Bluetooth connection to a smartphone, where the device is paired and managed via the MobECG mobile application. Initially, personal and other necessary information are entered into the smartphone application; then, the user can forget that he or she is wearing the device. The application works reliably in the background, even when using the phone for calls or other applications. If desired, the user can monitor the heart rate on the meter display with a curve and calculate it on an ongoing basis. Finally, the measurements are collected on the phone and can be transmitted to the physician in two ways: (1) pressing the button, the user can prepare a PDF report and send it to the physician's e-mail address or (2) transfer the data via USB cable to the physician's computer, where he or she can closely monitor the entire recording using VisECG. The first method is useful in the case of a severe disorder in which it is necessary to inform the physician. However, it is still related to the availability and responsiveness of the physician. When reading the recording, one should remember that it is not any standard lead typically used in a Holter monitor and that it is a single-channel measurement that is performed live on a patient moving and performing daily activities. The recordings can show different disorders but need to be evaluated so that artefacts can be distinguished from the actual disturbance of the rhythm. VisECG enables us to review and accurately analyze the recording and produce a report that can be submitted to physicians of other specialities for consultation or delivered to the patient and his or her physician as a measurement result. Given that the measurement is only a single channel, we can estimate the frequency and possible disturbances of rhythm but not ischemia.The study included the patients and their family physician. Patients with a complaint of heart rhythm disorder but no detectable rhythm disturbance on a 12-channel ECG record performed at the first visit were included. If a rhythm disturbance was detected at that time, the patient was treated according to the guidelines and was not included in the study. However, if a diagnosis of rhythm disorder could not have been made, the patient was included in the study. In the study, the investigators divided participants into two groups: test group where they received the personal ECG sensor and control group without the sensor one after another according to their visits at the office. However, the protocol was not followed rigorously, and physicians had the option of deciding for themselves if they prefer not to include the patient in the test group. The test group received an ECG sensor, which was placed by a healthcare professional and worn for three days. Whereat that time, they received information about the placement and handling of the sensor. The sensor was placed using two self-adhesive electrodes on the skin of the chest, which should not be too hairy. Then, the sensor was attached to the electrode and connected via Bluetooth to the smartphone, which was also provided to the patient with the charger for the duration of the examination. Patients were advised to perform their daily activities as regularly as possible and not to remove the sensor while showering or sleeping and keep the smartphone in the same room with them. In case the electrode peeled off, the patient had four spare electrodes and could install them himself. During the investigation, the patient kept a journal where he or she wrote down his or her problems and feelings. After 3 days, the patient returned to the healthcare provider, who removed the sensor and downloaded the measurements from the phone, which are then sent to the physicians who will analyze the reading. Then, the measurement was transferred to the computer memory and sent to the physicians for evaluation. The same patient underwent a checkup with the physician after 5-10 days, which depended on the date they had made an appointment. The physician read the recording, and in case of severe rhythm disorder, the patient was called earlier for a checkup at the physician's clinic where he or she received treatment as needed. The control group received a questionnaire and returned to the physician after 5-10 days.

For the purpose of the study, a questionnaire was made, and it was validated in a similar pilot study in a hospital setting. At the first visit to the doctor's office, all patients received a questionnaire to record their problems and provide an opinion on the quality and usefulness of the examination. Also, physicians of all tested patient had to complete two questionnaires. One for a patient on the first visit, then after 5-10 days, and after 3 months. The questionnaire provided us with demographics data, chronic illness and medication, presence of possible rhythm disorder and actions taken after first and second visit. The other questionnaire was used to record their comments on the quality and usefulness of this method.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years,
* there was a history of suspected arrhythmia,
* at the time of examination, the ECG is within normal limits
* the patient has never been treated for any heart rhythm disorder.

Exclusion Criteria:

* age less than 18 years,
* on examination on the ECG, the patient was not in sinus rhythm, and
* that the patient has a known heart rhythm disorder and / or is being treated for it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who come to their family physician with the complaint of hearth rhythm disorder as selected time. Their family physicians are also included.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change from no detected hearth rhythm disorders to diagnosed hearth rhythm disorders at day 90 | baseline and day 90
  With the help of ECG sensor finding arrhythmias in patients where standard ECG record was normal. Change = (day 90 record - baseline record)

SECONDARY OUTCOMES:
Change in patients and doctors satisfaction with this method after detecting possible hearth rhythm disorders | baseline and day 90
  With the help of a questionnaire see how users are satisfied with this method after 3 months. Change = (day 90 record - baseline record)

CONTACTS AND LOCATIONS:
Overall Officials: Stasa Vodicka, MD, Principal Investigator — Health care center Murska Sobota
Locations (1):
- Health care center Murska Sobota, Murska Sobota, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mistry H. Systematic review of studies of the cost-effectiveness of telemedicine and telecare. Changes in the economic evidence over twenty years. J Telemed Telecare. 2012 Jan;18(1):1-6. doi: 10.1258/jtt.2011.110505. Epub 2011 Nov 18. PMID 22101609
- [Result] Lieberman J. How telemedicine is aiding prompt ECG diagnosis in primary care. Br J Community Nurs. 2008 Mar;13(3):123-6. doi: 10.12968/bjcn.2008.13.3.28676. PMID 18557568
- [Result] Orchard J, Freedman SB, Lowres N, Peiris D, Neubeck L. iPhone ECG screening by practice nurses and receptionists for atrial fibrillation in general practice: the GP-SEARCH qualitative pilot study. Aust Fam Physician. 2014 May;43(5):315-9. PMID 24791776
- [Result] Klein-Wiele O, Faghih M, Dreesen S, Urbien R, Abdelghafor M, Kara K, Schulte-Hermes M, Garmer M, Gronemeyer D, Hailer B. A novel cross-sector telemedical approach to detect arrhythmia in primary care patients with palpitations using a patient-activated event recorder. Cardiol J. 2016;23(4):422-8. doi: 10.5603/CJ.a2016.0033. Epub 2016 Jun 20. PMID 27320955
- See also: Use of personal digital ECG sensor — http://www.savvy.si

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT04463524/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT04463524/ICF_001.pdf